CLINICAL TRIAL: NCT05544552
Title: A Multicenter, Open-label Phase 1/2 Study of TYRA300 in Advanced Urothelial Carcinoma and Other Solid Tumors With Activating FGFR3 Gene Alterations (SURF301)
Brief Title: Safety and Preliminary Anti-Tumor Activity of TYRA-300 in Advanced Urothelial Carcinoma and Other Solid Tumors With FGFR3 Gene Alterations
Acronym: SURF301
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYR300-101
Record Dates: First submitted 2022-09-06; First posted 2022-09-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Solid Tumor; Urothelial Carcinoma; Solid Tumor, Adult; Bladder Cancer; Non-muscle-invasive Bladder Cancer; FGFR3 Gene Mutation; FGFR3 Gene Alteration; Advanced Solid Tumor; Advanced Urothelial Carcinoma; Urinary Tract Cancer; Urinary Tract Tumor; Urinary Tract Carcinoma
Keywords: bladder; FGFR3 gene activation; FGFR3 gene alterations; FGFR3 gene fusion/rearrangement; FGFR3 gene mutation; FGFR3 gene translocation; FGFR3 positive; Fibroblast growth factor receptor 3 (FGFR3); Fibroblast growth factor receptor 3 alterations; locally advanced cancer; metastatic cancer; solid tumors; urothelial cancer; urothelial carcinoma; Urinary tract cancer; Urinary tract tumor; Urinary tract carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Urologic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Part A - dose escalation (Experimental): TYRA-300 taken once daily by mouth in 28-day cycles starting at 10 mg daily.
  Interventions: Drug: TYRA-300
- Phase 1 Part B - dose expansion (Experimental): TYRA-300 taken once or twice daily by mouth in 28-day cycles.
  Interventions: Drug: TYRA-300
- Phase 2 (Experimental): TYRA-300 taken once or twice daily by mouth in 28-day cycles at doses determined during Phase 1.
  Interventions: Drug: TYRA-300

INTERVENTIONS:
Drug: TYRA-300 — TYRA-300 is an oral, novel potent FGFR 3-selective tyrosine kinase inhibitor that targets tumors that contain activating gene alterations of FGFR3.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of TYRA-300 in cancers with FGFR3 activating gene alterations, including locally advanced/metastatic urothelial carcinoma of the bladder and urinary tract and other advanced solid tumors.

DETAILED DESCRIPTION:
This is a single arm, multi-part, phase 1/2 global trial studying TYRA-300, a novel, potent fibroblast growth factor receptor (FGFR) 3-selective tyrosine kinase inhibitor, in advanced/metastatic urothelial carcinoma of the bladder and urinary tract, that contain activating gene alterations of FGFR3. Phase 1 is a dose-escalation study to evaluate the safety, tolerability, and PK of TYRA-300 to determine the optimal and maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). Phase 2 will evaluate the preliminary antitumor activity of TYRA-300 in cancers with FGFR3 activating gene alterations, including locally advanced/metastatic urothelial carcinoma of the bladder and urinary tract and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Part A and Part B

* Men and women 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
* Histologically confirmed advanced solid tumor who have exhausted standard therapeutic options.
* Evaluable (Part A) or measurable (Part B) disease according to RECIST v1.1.
* Histologically confirmed advanced solid tumor with an eligible FGFR3 gene mutation or fusion (Part B).

Phase 2

* Men and women 18 years of age or older.
* ECOG performance status of 0-2 or Karnofsky Performance Scale (KPS) >70.
* At least 1 measurable lesion by RECIST v1.1.
* Histologically confirmed locally advanced/metastatic tumor in one of the following categories:

  * Urothelial carcinoma with an eligible FGFR3 gene mutation or rearrangement who have progressed on a prior FGFR inhibitor and presence of a resistance mutation or other kinase domain mutation.
  * Urothelial carcinoma with an eligible FGFR3 gene mutation or rearrangement who has not received a prior FGFR inhibitor.
  * Any solid tumor with an eligible FGFR3 gene mutation or rearrangement.

Exclusion Criteria (All Phases):

* Has a serum phosphorus level > upper limit of normal (ULN) during screening that remains >ULN despite medical management.
* Any ocular condition likely to increase the risk of eye toxicity.
* History of or current uncontrolled cardiovascular disease.
* Active, symptomatic, or untreated brain metastases.
* Gastrointestinal disorders that will affect oral administration or absorption of TYRA-300.
* Females who are pregnant, breastfeeding, or planning to become pregnant and males who plan to father a child while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Part A: To determine the maximum tolerated doses (MTD). | Initiation of study treatment through 28 days.
Phase 1 Part B: To determine the recommended Phase 2 dose (R2PD). | Initiation of study treatment through 28 days (up to approximately 18 months).
Phase 2: Overall Response Rate (ORR), defined by RECIST v1.1. | Initiation of study treatment until disease progression, death, unacceptable toxicity, or withdrawal (up to 2 years).

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) as a measure of safety and tolerability. | Initiation of study treatment through 28-days post treatment (up to 2 years).
Frequency in changes in laboratory parameters and physical signs of toxicity. | Initiation of study treatment through 28-days post treatment (up to 2 years).
Pharmacokinetics: maximum plasma concentration (Cmax). | Initiation of study treatment through Cycle 3 Day 1 (each cycle is 28 days).
Pharmacokinetics: time to reach maximum plasma concentration (Tmax). | Initiation of study treatment through Cycle 3 Day 1(each cycle is 28 days).
Pharmacokinetics: area under the plasma concentration-time curve (AUC). | Initiation of study treatment through Cycle 3 Day 1 (each cycle is 28 days).
Pharmacokinetics: half-life of TYRA-300 (t1/2). | Initiation of study treatment through Cycle 3 Day 1 (each cycle is 28 days).
ORR is defined as the proportion of participants with complete response (CR) or partial response (PR) as determined by the investigator using RECIST V1.1. | From enrollment, every 8 or 12 weeks (up to 2 years).
Duration of response will be defined as the time from the initial CR or PR to the time of relapse or death, whichever occurs first among participant with an objective response. | From enrollment, every 8 or 12 weeks (up to 5 years).
Disease control rate is defined as the proportion of participants having a CR, PR or stable disease (SD) for >12 weeks. | From enrollment up to 5 years.
Time to response is defined as time to first CR or PR that is subsequently confirmed according to RECIST v1.1. | Up to 5 years.
Progression-free survival is defined as the time from the date of first study drug administration to the earliest date of documented disease progression or death. | From the date of the first dose of study drug until disease progression or death as assessed up to the last efficacy assessment for disease progression (up to 5 years)].

CONTACTS AND LOCATIONS:
Overall Officials: Doug Warner, Study Chair — Tyra Biosciences, Inc
Locations (19):
- United States (7):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center, Worchester, Massachusetts
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - Duke Cancer Institute (DCI) - Duke Cancer Center, Durham, North Carolina
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Vanderbilt University Medical Center (VUMC) - Vanderbilt-Ingram Cancer Center (VICC) - Nashville, Nashville, Tennessee
  - Seattle Cancer Care Alliance (SCCA) - South Lake Union, Seattle, Washington
- Australia (6):
  - Macquarie University, Macquarie Park, New South Wales
  - Tasman Oncology, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Research Unit, Melbourne, Victoria
  - Linear Clinical Research Limited, Nedlands, Washington
- France (3):
  - Institut de Cancerologie de L'Ouest (ICO), Saint-Herblain
  - Institut Claudius Regaud, IUCT-Oncopole, Toulouse
  - Gustave Roussy (Institut de Cancerologie Gustave-Roussy), Villejuif
- Spain (3):
  - NEXT Barcelona - Hospital Quironsalud Barcelona, Barcelona
  - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona
  - NEXT Madrid - Hospital Universitario Quironsalud Madrid, Madrid